CLINICAL TRIAL: NCT05941169
Title: A Prospective Study of Primary Metastatic Renal Cell Carcinoma Treated With Immunecheckpoint Inhibitors and Cytoreductive Nephrectomy vs Primary Tumour in Place
Brief Title: Primary Metastatic Renal Cell Carcinoma Treated With Immunecheckpoint Inhibitors and Cytoreductive Nephrectomy
Acronym: PrimerX
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Comprehensive Cancer Centre The Netherlands (Other)
Responsible Party: Principal Investigator, Adriaan D. Bins, Principal Investigator, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 83948
Record Dates: First submitted 2023-06-22; First posted 2023-07-12 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-07

CONDITIONS: Renal Cell Carcinoma
Keywords: Cytoreductive Nephrectomy; Immunotherapy; Tyrosine Kinase Inhibitor
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cytoreductive Nephrectomy (Experimental): Cytoreductive Nephrectomy within 6 months to 1 year after start systemic therapy for metastatic Renal Cell Carcinoma
  Interventions: Procedure: Cytoreductive Nephrectomy
- Standard of Care (No Intervention): Standard of Care for metastatic Renal Cell Carcinoma

INTERVENTIONS:
Procedure: Cytoreductive Nephrectomy — The experimental intervention consists of cytoreductive nephrectomy (CN) or any ablative local therapy within 6 months and 1 year after start of systemic treatment. All types of ablative local therapy are allowed as a substitute for CN
  Arms: Cytoreductive Nephrectomy

SUMMARY:
The benefit of deferred Cytoreductive Nephrectomy (CN) has to be re-assessed in the context of IO +IO and IO + TKI systemic treatment. Given the benefit of CN in the setting of first generation immunotherapy, it is conceivable that both trials underestimated the benefit of CN, in absence of immunotherapy.

DETAILED DESCRIPTION:
In past years, much research has been done into the beneficial effects of cytoreductive nephrectomy in patients with metastatic renal cancer receiving systemic therapy with positive results. In the meantime systhemic therapy, and in particular immunotherapy, have changed. Patients with metastatic renal cancer are increasingly treated with immunocheckpoint inhibitors, but the effect of adding cytoreductive nephrectomy in this group of patients has not yet been investigated. The aim of this study is to investigate whether performing a cytoreductive nephrectomy has a beneficial effect on overall survival in patients with metastatic renal cancer receiving systemic therapy using immunocheckpoint inhibitors.

A randomized controlled trial. All eligible patients have already been enrolled in the PRO-RCC registry, a registry that collects prospective observational data, and have also given consent to be included in other studies as a control cohort. This design is called a TWiC (trial within cohort). After randomization, patients who are randomized into the therapy arm will receive a patient information via their treating physician. Upon participation, an informed consent will be signed and the patient will be scheduled for surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients age ≥ 18 years
2. Signed and written informed consent Note: Written and signed informed consent will be obtained before any study procedures, including study-specific-screening procedures, has been performed.
3. Informed consent obtained for being offered future experimental interventions within the PRO-RCC project.
4. Histologically confirmed diagnosis of metastatic clear cell, papillary or chromophobe renal cell carcinoma of intermediate to poor risk, including sarcomatoid features, with
5. World Health Organization (WHO) performance status of 0-1.
6. Surgical candidates based on surgeon and anesthetist assessment
7. Treatment with an IO combination (IO+IO or IO+TKI) as standard of care for metastatic RCC
8. Absence of progression at metastatic sites at time of identification (6month after start of systemic first line treatment). 9) Primary tumor in situ 10) Participation in the PRO-RCC prospective cohort.

Exclusion Criteria:

NA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 750 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2030-04-01 (Estimated); Study Completion 2031-04-01 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | defined as time from randomization to death of any cause during 5 years of follow-up
  Overall Survival Using Kaplan Meier Survival analysis

SECONDARY OUTCOMES:
Long term Quality of Life outcomes using validated EORTC Quality of Life Questionnaire (QLQ-C30) | Post operative follow-up period during 5 years
  using the Dutch validated EORTC Quality of Life Questionnaire (QLQ-C30)
Surgical morbidity outcomes using Clavien Dindo classification of surgical morbidity | Post operative follow-up period during 5 years
  Clavien Dindo classification of surgical morbidity is used to classify morbidity outcomes

OTHER OUTCOMES:
Clinical data and annotated tissue for translational research into mechanisms of treatment response and resistance. | post-operative follow-up period during 5 years
  In detail, we will examine the intratumor alteration of tumor infiltrating CD8, CD4, NK(T) cells (CD56+,CD3+-), and the distribution of these NK cells in the tumor, as these cells have been shown to be involved in anti-tumor responses in RCC.

CONTACTS AND LOCATIONS:
Overall Officials: Adriaan Bins, MD PhD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Figaroa O, Zondervan P, Kessels R, Berkhof J, Aarts M, Hamberg P, Los M, Piersma D, Rikhof B, Suelmann B, Tascilar M, van der Veldt A, Verhagen P, Westgeest H, Yildirim H, Bex A, Bins A. PrimerX: A Bayesian Multistage Cohort Embedded Randomised Trial to Evaluate the Role of Deferred Local Therapy of the Primary Tumour in Combination with Immune Checkpoint Inhibitor-based First-line Therapy in Metastatic Renal Cell Carcinoma Patients. Eur Urol Open Sci. 2024 Oct 14;70:28-35. doi: 10.1016/j.euros.2024.09.002. eCollection 2024 Dec. PMID 39483517